CLINICAL TRIAL: NCT05049031
Title: Study of the Impact of Adjuvant Hormone Therapy on Bone and Cardiovascular Risk After Initial Treatment in Patients With Non-metastatic Breast Cancer
Brief Title: Impact of Adjuvant Hormone Therapy on Bone and Cardiovascular Risk
Acronym: IMPACTTHKS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC31/21/0368
Record Dates: First submitted 2021-09-09; First posted 2021-09-17 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast cancer treated with hormone therapy (Experimental): Adult patients with T1-T3, N0-N2, M0 breast cancer and referred to the Menopause Center of Toulouse Hospital for their breast cancer
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A questionnaire will be given to patients who will ask them about their possible fractures, their bone and oncological follow-ups and their possible cardiovascular events since the end of treatment with hormone therapy.

SUMMARY:
Breast cancer is the most frequently observed cancer in women in France.The mortality rate is still decreasing with a decrease of 1.6% per year between 2010 and 2018, explained by the improvement in available treatments.For patients with breast cancer expressing hormone receptors, treatment with Tamoxifen or anti-aromatase can have the risk of the cancer coming back.However, these treatments have many side effects, including the risk of osteoporosis and metabolic disorders with anti-aromatases; and arterial and thromboembolic accidents with Tamoxifen.These effects have been well studied while taking hormone therapy.However, very few studies have analyzed the impact of these treatments after stopping them in women who have had non-metastatic hormone-sensitive breast cancer and uncertainties persist on the evolution of the health risk after initial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who had T1-T3, N0-N2, M0 breast cancer
* Patients referred to the Menopause center in the context of their breast cancer who were included in the original study evaluating the bone impact of hormone therapy carried out between 2010 "Bone and cardiovascular impact of adjuvant hormone therapy for cancer non-metastatic breast "
* Patient who has given her consent for the study (written or verbal) after clear and fair information

Exclusion Criteria:

* Metastatic breast tumor
* Absence of adjuvant hormone therapy for patients whose tumor did not express hormone receptors
* Patients who have died since the last assessment
* Protected adult patient (guardianship, curatorship, safeguard of justice)

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the bone impact of hormone therapy remotely | Inclusion day (day 0)
  A questionnaire asking patients if they have fractures since stopping the treatment will be offered.
Evaluate the cardiovascular impact of hormone therapy remotely | Inclusion day (day 0)
  A questionnaire asking patients if they have had a cardiovascular problem since stopping treatment will be offered.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Gosset, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No